CLINICAL TRIAL: NCT06813131
Title: The Effect of Medical Nutrition Therapy and Follow-Up Frequency on Parameters Related to Metabolic Syndrome in Individuals With Metabolic Syndrome: A Randomized Controlled Trial
Brief Title: Impact of Medical Nutrition Therapy and Follow-Up Frequency on Metabolic Syndrome Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kubra Yildiz Guler, Research University, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HU-BVD-KYG-01
Record Dates: First submitted 2025-01-28; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Metabolic Syndrome; Metabolic Syndrome Obesity; Metabolic Syndrome Parameters
Keywords: metabolic syndrome x; abdominal obesity; medical nutrition therapy
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Abdominal | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Three groups: Intervention group, Intensive intervention group, Control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Group (Experimental): Participants in this group attended face-to-face consultations at baseline, and at the 1st, 2nd, and 3rd months (a total of four visits). These sessions focused on providing guidance for dietary and lifestyle modifications.
  Interventions: Other: Dietary counseling; Other: calling via telephone
- Intensive Intervention (Experimental): This group followed the same face-to-face consultation schedule as the intervention group (baseline, 1st, 2nd, and 3rd months). In addition, participants were contacted weekly via phone to assess dietary adherence and provide ongoing motivation and support, making this a more frequent and intensive intervention.
  Across all groups, the study primarily aimed to evaluate changes in weight loss, blood sugar, lipid levels, and metabolic syndrome parameters, while assessing the impact of intervention intensity on these outcomes.
  Interventions: Other: Dietary counseling
- Control Group (No Intervention): Participants in this group were seen in person only twice, at baseline and at the 3rd month. No additional interventions were applied, and the aim was to observe the natural course of their condition.

INTERVENTIONS:
Other: Dietary counseling — This intervention uniquely focuses on the frequency of dietitian-led follow-up visits and their impact on metabolic syndrome-related parameters. The study includes three distinct groups with varying levels of follow-up intensity (control, intervention, and intensive intervention).
  Arms: Intensive Intervention; Intervention Group
Other: calling via telephone — The intensive intervention group involves weekly diet adherence assessments via phone calls, setting it apart from other studies that typically rely on less frequent or standardized follow-up schedules. This design allows for the evaluation of how consultation frequency influences outcomes such as weight loss, blood sugar levels, lipid profile, and metabolic syndrome components."
  Arms: Intervention Group

SUMMARY:
There is no study that has investigated the effects of medical nutrition therapy and more frequent follow-up via telehealth on metabolic syndrome parameters in patients with MetS who have multiple metabolic disorders such as being overweight, prediabetic/diabetic, dyslipidemic and having increased blood pressure. This study was conducted to examine the effects of medical nutrition therapy and increased follow-up via telephone calls on MetS-related parameters in individuals with MetS.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with HbA1c values <8.5%
* Diagnosed with MetS by a physician according to the criteria declared by the consensus of the "International Diabetes Federation Task Force on Epidemiology and Prevention, National Heart, Lung, and Blood Institute, American Heart Association, World Heart Federation, International Atherosclerosis Society, and International Association for the Study of Obesity" were included.

Exclusion Criteria:

* Taking anti diabetic agents other then metformin
* Taking anti hyperlipidemic agents
* Taking anti hypertensive agents
* Using food supplements (w-3, chromium, multivitamins) that could affect metabolic parameters,
* Having kidney failure,
* Having liver failure,
* Having immune failure
* Having chronic gastrointestinal system disease
* Having cancer
* Having type 1 diabetes
* Being pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-10-14 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
waist circumference | Baseline, 1 month, 2 months, and 3 months after the start of the intervention
  Waist circumference, which is an indicator of abdominal obesity, the central component of metabolic syndrome, was determined as the primary outcome because of its strong association with cardiometabolic risk and its correlation with other MetS components, and because it is a significant measure in reflecting the overall effect of the intervention.

SECONDARY OUTCOMES:
fasting plasma glucose, triglyceride, HDL-C and blood pressure (Number of metabolic syndrome criteria) | Baseline, 1 month, 2 months, and 3 months after the start of the intervention
  The change in the number of individuals with the following metabolic syndrome criteria has been determined as a secondary outcome:
  * Elevated fasting plasma glucose (number of individuals with ≥100 mg/dL),
  * Elevated triglycerides (number of individuals with ≥150 mg/dL),
  * Low HDL-C (number of individuals with <50 mg/dL in women and <40 mg/dL in men),
  * Elevated blood pressure (number of individuals with systolic ≥130 mmHg and/or diastolic ≥85 mmHg).
  Multiple assessments with different units of measurement will be combined into a single reported value based on the change in the number of individuals meeting these conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul, Kadıkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF

REFERENCES:
- [Background] Zujko ME, Rozniata M, Zujko K. Individual Diet Modification Reduces the Metabolic Syndrome in Patients Before Pharmacological Treatment. Nutrients. 2021 Jun 19;13(6):2102. doi: 10.3390/nu13062102. PMID 34205362
- [Background] Alfawaz HA, Wani K, Alnaami AM, Al-Saleh Y, Aljohani NJ, Al-Attas OS, Alokail MS, Kumar S, Al-Daghri NM. Effects of Different Dietary and Lifestyle Modification Therapies on Metabolic Syndrome in Prediabetic Arab Patients: A 12-Month Longitudinal Study. Nutrients. 2018 Mar 20;10(3):383. doi: 10.3390/nu10030383. PMID 29558423
- [Background] Parker AR, Byham-Gray L, Denmark R, Winkle PJ. The effect of medical nutrition therapy by a registered dietitian nutritionist in patients with prediabetes participating in a randomized controlled clinical research trial. J Acad Nutr Diet. 2014 Nov;114(11):1739-48. doi: 10.1016/j.jand.2014.07.020. Epub 2014 Sep 11. PMID 25218597